CLINICAL TRIAL: NCT01283633
Title: Investigation of the Use of Remote Presence Robots in the Administration of Neuromodulation Treatment
Brief Title: Investigation of the Use of Remote Presence Robots in Delivery of Neuromodulation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Ivar Mendez, Neurosurgeon, Nova Scotia Health Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Robotics-Neuromod-Mendez
Record Dates: First submitted 2011-01-18; First posted 2011-01-26 (Estimated); Last update posted 2012-03-12 (Estimated); Status verified 2012-03

CONDITIONS: Complications; Neurostimulator; Satisfaction
Keywords: neuromodulation; remote presence robotics
MeSH Terms: conditions — Personal Satisfaction | interventions — Transcutaneous Electric Nerve Stimulation; Deep Brain Stimulation; Spinal Cord Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- programming with non-experienced nurse (Experimental): Programming done by an experienced neuromodulation clinician will be compared to the patient satisfaction of a programming session with an inexperienced nurse via remote presence robotics, which will be directed by the experienced clinician
  Interventions: Device: Neuromodulation

INTERVENTIONS:
Device: Neuromodulation — Neuromodulation as directed via remote presence robotic and experienced clinician for those with neuromodulation systems implanted to treat movement disorders and chronic pain
  Other Names: Neurostimulation; deep brain stimulation; spinal cord stimulation

SUMMARY:
In recent years, robotic devices are becoming more and more common in medical practice. Such devices provide an effective way to communicate within a clinical setting, but recent studies have shown far more diverse uses for these robots, ranging from training future surgeons to diagnoses of patients. In the investigators study, the investigators would like to investigate whether it is effective to employ robotic devices in the administration of neurostimulation treatment. It is the investigators hypothesis that the introduction of robotic devices will only yield minimal if any inaccuracies in a standard neuromodulation treatment protocol. In addition, the investigators also predict a high satisfaction rating from all participants involved in conditions involving the robot.

DETAILED DESCRIPTION:
Patients with neuromodulation systems implanted for either movement disorders or chronic pain and who require programming of their systems will be approached to enter the study. Those who consent will be consecutively assigned to either the normal standard of care (i.e. programming of their systems with an experienced clinician) or programming of their systems with an inexperienced programmer (nurse) who will be directed by the experienced programmer via the remote presence robot. Both the nurses and the patients will complete questionnaires rating their satisfaction of the programming experience.

They will each only receive one questionnaire at the end of the programming session. There is no other test point.

ELIGIBILITY:
Inclusion Criteria:

* patients with neuromodulation systems, requiring programming
* nurses who have never programmed a neuromodulation system before

Exclusion Criteria:

* those who are unwilling to give consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction | Patients will complete the questionnaire once following the neuromodulation therapy. Day 1
  The questionnaire will take approximately 10 minutes to complete. There are no other follow-ups required. This is the only study time commitment for the patients above the usual standard of care.

SECONDARY OUTCOMES:
Nursing satisfaction questionnaire | Immediately following the neuromodulation session, the nurse will complete one questionnnaire. Day 1.
  The questionnaire will take approximately 10 minutes to complete. The time commitment from the nurse programmer will be approximately 45 minutes. There are no other test points nor follow up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Ivar M Mendez, MD, Principal Investigator — Capital Health and Dalhousie University
Locations (1):
- Centre for Clinical Research, Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia, Canada